CLINICAL TRIAL: NCT01470300
Title: Reducing Energy Density by Different Methods to Decrease Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Principle Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FoodED401; R37DK039177-19 (NIH); 2R01DK059853-10 (NIH)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard ED (Experimental): 100% energy density
  Interventions: Other: Energy density feeding study
- Reduced ED - F/V (Experimental): 80% energy density by adding fruit and vegetables
  Interventions: Other: Energy density feeding study
- Reduced ED - Fat (Experimental): 80% energy density by decreasing fat
  Interventions: Other: Energy density feeding study
- Reduced ED - Plain water (Experimental): 80% energy density by adding plain water
  Interventions: Other: Energy density feeding study

INTERVENTIONS:
Other: Energy density feeding study — In a crossover design, adults are served breakfast, lunch, and dinner, 1 day a week for 4 weeks. Meal entrees will vary in energy density (100% and 80%) and the method used to reduce the energy density (added fruit & vegetables, decreased fat, added plain water).

SUMMARY:
The purpose of this research is to investigate how using different methods to reduce the energy density of entrees affects daily energy intake in adults. It is hypothesized that reducing the energy density of entrees will decrease energy intake. It is also hypothesized that reducing the energy density by incorporating fruit and vegetables will decrease energy intake more than reducing the energy density by decreasing fat content or adding plain water.

ELIGIBILITY:
Inclusion Criteria:

* Adults from Penn State and surrounding community

Exclusion Criteria:

* Currently dieting
* Food allergies

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Energy intake | 1 month

SECONDARY OUTCOMES:
Food intake | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States